CLINICAL TRIAL: NCT01616108
Title: Bupivacaine Injection of Eye Muscles to Treat Strabismus
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Smith-Kettlewell Eye Research Institute (Other)
Collaborators: Eidactics (Other); Sutter Health (Other); Strabismus Research Foundation (Other)
Responsible Party: Principal Investigator, Alan B. Scott, Senior Scientist, Smith-Kettlewell Eye Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPX-STRAB
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Strabismus; Esotropia; Exotropia; Graves Disease; Ptosis, Eyelid
Keywords: strabismus; diplopia
MeSH Terms: conditions — Strabismus; Esotropia; Exotropia; Graves Disease; Blepharoptosis; Diplopia | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bupivacaine Injection (Experimental): Differences in concentration from 0.75% to 3.0% are compared. Differences in volume for 1.0 mL to 3.0 mL are compared. Differences in compounding with addition of epinephrine will be used and compared to plain bupivacaine.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Differences in concentration from 0.75% to 3.0% are compared. Differences in volume for 1.0 mL to 3.0 mL are compared. Differences in compounding with addition of epinephrine will be used and compared to plain bupivacaine.
  Other Names: Marcaine

SUMMARY:
This study seeks to determine if bupivacaine injection of eye muscles can make them stronger and stiffer, and thereby correct the position of eyes that are turned in or mis-aligned, a condition generally termed strabismus. It seeks further to find out the different effects of various concentrations or formulations of bupivacaine, and whether addition of Botox to other eye muscles can add to the effect of bupivacaine and enhance the correction of strabismus.

DETAILED DESCRIPTION:
Patients eligible for inclusion in the study will be age 8 to 95 years and have an eye deviation (strabismus) that is potentially subject to surgical correction.

The eye alignment will be measured. The eye muscles may be measured by MRI. The eye will be anesthetized by eye drops. One or more eye muscles will be injected with bupivacaine. Botox® will be injected into the antagonist muscle in some cases to increase the effect of the bupivacaine.

Data on the strabismus deviation, any side effects of the drug injection, and the eye muscles as measured by MRI, will be recorded at intervals after injection. These data will be compared with the like measurements taken before injection.

The primary outcome will be the eye alignment change at 180 days. A secondary outcome will be the change in muscle size, strength, or stiffness.

For large strabismus deviations not fully corrected by a first injection, a second injection can be made. Follow-up alignment and muscle measurements will be as for the initial injection.

ELIGIBILITY:
Inclusion Criteria:

* Clinical pattern of strabismus of 5 prism diopters or more

Exclusion Criteria:

* Active eye infection

Ages: 8 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-04; Primary Completion 2019-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Eye alignment | 6 months after injection
  Alignment of the two eyes as measured by prism cover test or other applicable test

SECONDARY OUTCOMES:
Percentage correction of the pre-treatment eye deviation | 6 months after injection treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alan B Scott, MD, Principal Investigator — Strabismus Research Foundation; Joel M Miller, PhD, Principal Investigator — Strabismus Research Foundation
Locations (1):
- Strabismus Research Foundation, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller JM, Scott AB, Danh KK, Strasser D, Sane M. Bupivacaine injection remodels extraocular muscles and corrects comitant strabismus. Ophthalmology. 2013 Dec;120(12):2733-2740. doi: 10.1016/j.ophtha.2013.06.003. Epub 2013 Aug 2. PMID 23916485
- [Background] Scott AB, Miller JM, Shieh KR. Bupivacaine injection of the lateral rectus muscle to treat esotropia. J AAPOS. 2009 Apr;13(2):119-22. doi: 10.1016/j.jaapos.2008.10.016. PMID 19393509
- [Background] Scott AB, Alexander DE, Miller JM. Bupivacaine injection of eye muscles to treat strabismus. Br J Ophthalmol. 2007 Feb;91(2):146-8. doi: 10.1136/bjo.2006.110619. Epub 2006 Nov 29. PMID 17135337
- [Background] Debert I, Miller JM, Danh KK, Scott AB. Pharmacologic injection treatment of comitant strabismus. J AAPOS. 2016 Apr;20(2):106-111.e2. doi: 10.1016/j.jaapos.2015.11.011. PMID 27079589
- [Result] Scott AB, Miller JM, Shieh KR. Treating strabismus by injecting the agonist muscle with bupivacaine and the antagonist with botulinum toxin. Trans Am Ophthalmol Soc. 2009 Dec;107:104-9. PMID 20126486
- See also: Homepage for The Strabismus Research Foundation. — http://www.srfsf.org